CLINICAL TRIAL: NCT00615277
Title: The Effect of Long-Chain Polyunsaturated Fatty Acids on Cognitive Performance and Mood of Healthy Young Adults
Brief Title: The Effect of Long-Chain Polyunsaturated Fatty Acids on Cognitive Performance and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Philipps University Marburg (Other); Cognitive Drug Research Ltd (Unknown)
Responsible Party: Prof. Dr. Dr. Manfred Spitzer, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 213/2005; 213/2005
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2008-02

CONDITIONS: Healthy
Keywords: Young adults; Long-chain polyunsaturated fatty acids; Cognitive function; Mood; Supply with omega-3 fatty acids
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1: omega-3 fatty acid supplement
  Interventions: Dietary Supplement: Omega-3 fatty acids
- 2 (Placebo Comparator): 2: olive oil
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — 600 mg EPA 120mg DHA daily, 16 weeks

SUMMARY:
The study investigates whether dietary intake of omega-3 long-chain polyunsaturated fatty acids affects learning and mood of healthy young adults.

DETAILED DESCRIPTION:
The long-chain polyunsaturated fatty acids (LCPUFA) EPA (eicosapentaenoic acid), DHA (docosahexaenoic acid) of the omega-3 series and AA (arachidonic acid) of the omega-6 series are building blocks of all cell membranes and are found in high concentrations in retina and brain. Food sources of LA and ALA are vegetable oils, nuts and seeds. Since low conversion rates from ALA to DHA are a characteristic of human metabolism, adequate dietary provision with the long-chained omega-3 molecules depends primarily on individual eating habits. While AA is abundant in meat and dairy products, EPA and DHA are found in noteworthy concentrations only in certain species of fatty fish, such as salmon or mackerel.

The study investigates whether participants receiving an omega-3 supplement over a period of 4 month, perform better on a series of cognitive tests, than the participants allocated to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults

Exclusion Criteria:

* Coagulation disorder

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2006-10; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cognition | Before intervention and after 16 weeks of intervention

SECONDARY OUTCOMES:
Mood | Before intervention and after 16 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katharina A Widenhorn-Mueller, PhD, Principal Investigator — University of Ulm; Ulrike Weiland, MD, Principal Investigator — University of Ulm